CLINICAL TRIAL: NCT02800343
Title: The Contribution of Intraoperative Mechanical Red Cell Salvage to Acidosis in the Immediate Postoperative Period After Cardiac Surgery
Brief Title: Intraoperative Cell Salvage and Postoperative Acidosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16077
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Acidosis
MeSH Terms: conditions — Acidosis | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiovascular surgery: All adult patients undergoing elective or emergency cardiovascular surgery at the study site
  Interventions: Procedure: routine administration of 0.9% sodium chloride

INTERVENTIONS:
Procedure: routine administration of 0.9% sodium chloride — 0.9% sodium chloride is used as the wash and suspension solution for red blood cells during the Intraoperative red blood cell salvage (ICS) procedure.
  Other Names: Baxter 0.9% sodium chloride

SUMMARY:
Metabolic acidosis is a common complication that patients experience in the early postoperative period following cardiac surgery. Increasingly, the composition and volume of intravenous fluids administered during surgery have been implicated in the development of postoperative acidosis. Intraoperative Cell Salvage (ICS), an autologous blood transfusion technique employed by Cardiac/Perfusion Units to minimize blood loss during surgery, involves the infusion of of one such fluid, 0.9% sodium chloride. The rapid infusion of large volumes of 0.9% sodium chloride has previously been linked with the development of hyperchloraemic acidosis. It was therefore hypothesized that the volume of mechanically salvaged of red blood cells re-infused into patients undergoing heart surgery contributes to the acidosis that occurs in the early postoperative period.

To test this, the investigators have designed an observational cohort study to check for correlation between the volume of cell salvaged blood infused during surgery and the severity of postoperative acidosis (which will be assessed using data from routine arterial blood gas samples).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients scheduled for cardiac surgery including both on- and off-pump coronary artery bypass grafting surgery, heart valve surgery, septal surgery, and aortic surgery)
* Patients must have consented to participate

Exclusion Criteria:

* Patients under 18 years of age
* Patients who are unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing elective or emergency cardiovascular surgery at the study site (Royal Infirmary of Edinburgh) during the data collection phase of the project will be approached for consent.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
plasma hydrogen ion concentration | at the start of surgery (before fluid infusion) and immediately after surgery (after fluid infusion)
  Plasma hydrogen ion concentration is measured by the arterial blood gas analyzer machine, and serves as a direct indicator of plasma acidity at a given time point.
  Data from two routine blood gas samples are of interest:
  T1 - baseline measurement taken on insertion of an arterial line immediately after the induction of anaesthesia (i.e. before any fluid infusion has commenced); T2 - postoperative measurement made immediately after patient arrives in ICU (i.e. once all the cell salvaged blood has been transfused)

SECONDARY OUTCOMES:
plasma chloride concentration | at the start of surgery (before fluid infusion) and immediately after surgery (after fluid infusion)
  Plasma chloride concentration is measured by the arterial blood gas analyzer machine.
  Data from two routine blood gas samples are of interest:
  T1 - baseline measurement taken on insertion of an arterial line immediately after the induction of anaesthesia (i.e. before any fluid infusion has commenced); T2 - postoperative measurement made immediately after patient arrives in ICU (i.e. once all the cell salvaged blood has been transfused)
plasma strong ion difference | at the start of surgery (before fluid infusion) and immediately after surgery (after fluid infusion)
  Plasma strong ion difference can be computed from routine arterial blood gas electrolyte measurements (chloride, lactate, sodium, potassium) using a formula.
  Strong ion difference serves as an indirect measure of plasma acidity.
  Data from two routine blood gas samples are of interest:
  T1 - baseline measurement taken on insertion of an arterial line immediately after the induction of anaesthesia (i.e. before any fluid infusion has commenced); T2 - postoperative measurement made immediately after patient arrives in ICU (i.e. once all the cell salvaged blood has been transfused)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Alston, MBChB, FRCA, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The findings of the study will be written up as a scientific report, which will be submitted for publication in a peer-reviewed scientific journal and presented at a conference.
  At the time of publication/dissemination, individual participant data will be reported as an aggregate.